CLINICAL TRIAL: NCT01359098
Title: Safety and Efficacy of Once-Daily Dosing of Ciprodexa Otic Foam (Ciprofloxacin 0.3% and Dexamethasone 0.1% Otic Foam) Compared to Twice-Daily Dosing of Ciprodex (0.3% Ciprofloxacin and Dexamethasone 0.1% Otic Suspension) in Patients With Acute Otitis Externa
Brief Title: Efficacy and Safety of Once-Daily Ciprodexa Otic Foam Compared to Twice-daily Ciprodex Ear Drops in Acute Otitis Externa
Acronym: Ciprodexa Foam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otic Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP-003-000
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Otitis Externa; Otorhinolaryngologic Diseases; Ear Diseases; Otitis
Keywords: swimmer's ear; ear drops; ear foam; otic foam; ear infection; ear pain; ear inflammation
MeSH Terms: conditions — Otitis Externa; Otorhinolaryngologic Diseases; Ear Diseases; Otitis; Earache | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciprodex Otic Suspension (Active Comparator): Ciprodex Sterile Otic Solution (Alcon, Inc.)
  Interventions: Drug: Ciprodex Otic Suspension
- Ciprodexa Otic Foam (Experimental): Ciprodexa Otic Foam (0.3% Ciprofloxacin, 0.1% Dexamethasone otic foam)
  Interventions: Drug: Ciprodexa Otic Foam

INTERVENTIONS:
Drug: Ciprodex Otic Suspension — 4 gtt b.i.d. for 7 days.
  Other Names: Ciprodex; Ciprodex b.i.d.
  Arms: Ciprodex Otic Suspension
Drug: Ciprodexa Otic Foam — 0.3% Ciprofloxacin, 0.1% Dexamethasone Otic Foam, 1 actuation, q.d. for 7 days
  Other Names: Ciprofloxacin, Dexamethasone Otic Foam; Ciprodexa foam once-a-day
  Arms: Ciprodexa Otic Foam

SUMMARY:
The purpose of this study is to assess the Safety and Efficacy of Ciprodexa Foam (0.3% Ciprofloxacin, 0.1% Dexamethasone Otic Foam), used once-a-day for 7 days for the treatment of Acute Diffuse Otitis Externa, compared to Ciprodex otic suspension used twice daily for 7 days.

DETAILED DESCRIPTION:
Acute otitis externa (AOE) is defined as a diffuse inflammation of the external ear canal, which may also involve the pinna and/or the tympanic membrane. AOE is one of the most common infections encountered by otolaryngologists, pediatricians and family physicians. Diagnosis of AOE requires rapid onset (generally within 48 hours) of symptoms and signs of ear canal inflammation which includes: A) otalgia (often severe), itching or fullness, sometimes accompanied by reduced hearing or jaw pain; B) tenderness of the tragus and/or pinna; and C) diffuse ear canal edema with or without erythema, sometimes accompanied by ear discharge (otorrhea).

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 years to 80 years old.
* Have a clinical diagnosis of Acute Otitis Externa based on clinical observation and of presumed bacterial origin.
* Intact tympanic membrane
* Unilateral disease

Exclusion Criteria:

* Known allergy or sensitivity to Ciprofloxacin or other quinolones.
* Clinical Diagnosis of chronic suppurative otitis media (CSOM), acute otitis media (AOM), involvement of middle ear effusion (MEE).
* Patient has the non intact tympanic membrane.
* Patient has a serious underlying disease.
* Patients with known history of immune dysfunction/deficiency and those receiving immunosuppressive therapy.
* Patients with history of Diabetes mellitus.
* Patients with more than 80% of the ear canal occluded.
* Pregnant or lactating patients.
* Overt fungal Acute Otitis Externa.
* Local ear canal abnormalities such as abscess, granulation or polyps.
* Congenital abnormalities of the external auditory canal or obstructive bony exostosis in the treated ear.
* Mastoid or other suppurative non-infectious ear disorder (e.g. cholesteatoma) in the treated ear.
* Seborrheic dermatitis or other dermatological conditions of the external auditory canal which would complicate evaluation.
* Current Infection requiring systemic antimicrobial therapy.
* Current or previous use of topical or oral antibiotics (within 3 days) or long-acting antibiotics (within 7 days).
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Clinical cure [lack of need of additional therapy] | Between Day 8 and Day 14 [e.g. 7 days after completion of treatment] that lasts 7 days
  Clinical cure [lack of need of additional therapy] confirmed by significant reduction or absence of the disease symptoms a) Otalgia/ear pain, b) tenderness with movement of pinna, c) edema/ear canal occlusion and d) ear discharge/otorrhea

SECONDARY OUTCOMES:
Otalgia/ear pain | At Visit 1, [Day 1 ,Baseline visit], at Visit 2 [Day 3 - Day 4, during treatment] and at Visit 3 Test-of-cure [Day 8 to Day 14]
  Ear pain as reported by the patient
Inflammation/ear edema | At the test-of-cure visit [Day 8 to Day 14]
Ear discharge/otorrhea | At the test-of-cure visit [Day 8 to Day 14]
tenderness with movement of pinna | At the test-of-cure visit [Day 8 - Day 14]

CONTACTS AND LOCATIONS:
Overall Officials: Yehudah Roth, MD, Principal Investigator — Edith Wolfson Medical Center
Locations (7):
- Israel (7):
  - Meir Medical Center, Kfar Saba, Israel
  - HaEmek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Wolfson Medical Center, Holon
  - Clalit Health Services - Raziel Clinic, Netanya
  - Maccabi Healthcare Services (H.M.O.), Tel Aviv
  - Sourasky Medical Center (Ichilov), Tel Aviv